CLINICAL TRIAL: NCT05884762
Title: earlY Upper Limb Rehabilitation WIth EEG-Neurofeedback After Stroke
Acronym: YUWIN-Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Fondation de l'Avenir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 35RC22_9743_YUWIN-Stroke; 2023-A01150-45 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-05-23; First posted 2023-06-01 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Stroke; Stroke Hemorrhagic; Stroke, Ischemic; Stroke Rehabilitation; Brain Infarction
Keywords: Stroke; Rehabilitation; neurofeedback; Upper Limb
MeSH Terms: conditions — Stroke; Hemorrhagic Stroke; Ischemic Stroke; Brain Infarction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The occupational therapist who will include and do the sessions will be open. The assessors who will test motor functions during the assessments will be blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): electroencephalographic neurofeedback + traditional reference rehabilitation programme
  Interventions: Other: electroencephalographic neurofeedback
- Control group (Sham Comparator): SHAM electroencephalographic neurofeedback + traditional reference rehabilitation programme
  Interventions: Other: SHAM electroencephalographic neurofeedback

INTERVENTIONS:
Other: electroencephalographic neurofeedback — The patient is installed in a quiet, isolated room in the Physical Medicine and Rehabilitation Department. The patient sits comfortably in front of a computer. A nurse or a rehabilitator installs the EEG headset and places gel in the electrodes (x32). Connecting the amplifier and interface. Checking the correct positioning and contact of the electrodes (impedance).
  * Calibration phase at rest.
  * Working phase: the sessions last 24 minutes. The patient will be asked to concentrate on the affected arm, and to imagine a movement of this arm, to feel the sensations, without any real movement of the arm.
    * In the Neurofeedback group, the patient will receive visual feedback of a virtual hand moving on a computer screen in front of him/her, depending on his/her brain activations. He will also receive haptic feedback (vibrations) in the flexor muscles of his wrist.
  Arms: Interventional group
Other: SHAM electroencephalographic neurofeedback — The patient is installed in a quiet, isolated room in the Physical Medicine and Rehabilitation Department. The patient sits comfortably in front of a computer. A nurse or a rehabilitator installs the EEG headset and places gel in the electrodes (x32). Connecting the amplifier and interface. Checking the correct positioning and contact of the electrodes (impedance).
  * Calibration phase at rest.
  * Working phase: the sessions last 24 minutes. The patient will be asked to concentrate on the affected arm, and to imagine a movement of this arm, to feel the sensations, without any real movement of the arm.
    * In the SHAM group, the visual feedback and haptic feedback are randomly generated
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate the effect of early rehabilitation treatment by electroencephalographic neurofeedback on upper limb motor function after stroke.

Researchers will compare :

Interventional group: electroencephalographic neurofeedback + traditional reference rehabilitation programme Control group: SHAM electroencephalographic neurofeedback + traditional reference rehabilitation programme

ELIGIBILITY:
Inclusion Criteria:

* Unilateral ischaemic or haemorrhagic stroke
* Adult (18-80 years), both sexes
* Stroke < 3 weeks
* Upper limb deficit defined by Shoulder Abduction Finger Extension score <5 on day 3 of stroke; i.e., patients predicted to have incomplete recovery
* No participation-limiting comprehension problems
* With or without homonymous lateral hemianopia; with or without visuospatial hemineglect
* Free, informed and written consent signed by the patient or a member of the patient's family (in the case of a patient who is able to understand the information and give consent but has motor difficulties resulting in an invalid signature).
* Affiliated to french social security

Exclusion Criteria:

* Ischemic or hemorrhagic brain stem and/or cerebellum involvement
* Multiple strokes
* Stroke < 1 week; in order not to be deleterious by starting active rehabilitation too early after immediate stroke
* Aphasia with major comprehension impairment
* Contraindication to MRI

  * pacemaker or implantable defibrillator,
  * neurosurgical clips,
  * cochlear implants,
  * intra-orbital or encephalic metallic foreign bodies,
  * stents placed less than 4 weeks ago and osteosynthesis devices placed less than 6 weeks ago,
  * claustrophobia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Measurement of motor impairment by the Fugl-Meyer Assesment - Upper Extremity | 28 days
  Measurement of motor impairment by the Fugl-Meyer Assesment - Upper Extremity

SECONDARY OUTCOMES:
Changes in ACTIVE RANGE OF MOTION (CxA) composite score | 28 days
  Changes in ACTIVE RANGE OF MOTION (CxA) composite score
Changes in ACTIVE RANGE OF MOTION (CxA) composite score | 3 months
  Changes in ACTIVE RANGE OF MOTION (CxA) composite score
Changes in Action Research Arm Test (ARAT) score | 28 days
  Changes in Action Research Arm Test (ARAT) score
Changes in Action Research Arm Test (ARAT) score | 3 months
  Changes in Action Research Arm Test (ARAT) score
Changes in force emitted (in kg) during a palmar grip (JAMAR) | 28 days
  Changes force emitted (in kg) during a palmar grip (JAMAR)
Changes in force emitted (in kg) during a palmar grip (JAMAR) | 3 months
  Changes force emitted (in kg) during a palmar grip (JAMAR)
Progression in Evaluation of the Motor activiy Log (MAL) | 28 days
  Progression in Evaluation of the Motor activiy Log (MAL)
Progression in Evaluation of the Motor activiy Log (MAL) | 3 months
  Progression in Evaluation of the Motor activiy Log (MAL)
Progression in The Composite Functional Independence Scale (MIF) | 28 days
  Progression in The Composite Functional Independence Scale (MIF)
Progression in The Composite Functional Independence Scale (MIF) | 3 months
  Progression in The Composite Functional Independence Scale (MIF)
Progression in The Stroke Impact Scale (SIS) | 28 days
  Progression in The Stroke Impact Scale (SIS)
Progression in The Stroke Impact Scale (SIS) | 3 months
  Progression in The Stroke Impact Scale (SIS)
Brain activity measured by electroencephalogram : improvement in cerebral activations in target zones | 28 days
  Brain activity measured by electroencephalogram : improvement in cerebral activations in target zones
Brain datas (fMRI activity and CST tractography) | 28 days
  Brain datas (fMRI activity and CST tractography)

CONTACTS AND LOCATIONS:
Overall Officials: Simon BUTET, MD, Principal Investigator — Rennes CHU
Locations (1):
- Rennes Chu, Rennes, France